CLINICAL TRIAL: NCT00310050
Title: A Phase I Dose-Escalating Study of Induction Gemcitabine/Pemetrexed Followed by Pemetrexed and Concurrent Upper Abdominal Radiation Therapy in Patients With Locally Advanced Pancreatic Cancer
Brief Title: Pemetrexed, Gemcitabine, and Radiation Therapy in Treating Patients With Locally Advanced Pancreatic Cancer
Status: Terminated | Phase: Phase 1 | Type: Interventional
Why Stopped: slow accrual
Sponsor: Wake Forest University Health Sciences (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CDR0000466320; CCCWFU-57103; LILLY-H3E-US-X031; CCCWFU-BG04-529
Record Dates: First submitted 2006-03-29; First posted 2006-04-03 (Estimated); Results first posted 2018-11-30 (Actual); Last update posted 2018-11-30 (Actual); Status verified 2018-11

CONDITIONS: Pancreatic Cancer
Keywords: stage II pancreatic cancer; stage III pancreatic cancer; stage IV pancreatic cancer
MeSH Terms: conditions — Pancreatic Neoplasms | interventions — Pemetrexed; Radiotherapy

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: Yes

ARMS (1):
- Pemetrexed in combination with concomitant radiotherapy (Experimental): Patients will receive Pemetrexed plus Radiotherapy.
  Interventions: Drug: pemetrexed disodium; Device: Radiotherapy

INTERVENTIONS:
Drug: pemetrexed disodium — 500 milligrams per meter squared day will be given during weeks 1, 3 and 5 of the radiation (3 total doses of Pemetrexed during the radiation therapy).
Device: Radiotherapy — During the chemoradiation, the radiotherapy will be administered in 1.8 Gy/fractions after completion of the Pemetrexed infusion, and continue daily (Monday through Friday) for 5 1/2 weeks for a total delivered dose of 50.4 Gy (Total of 28 radiation treatments).

SUMMARY:
RATIONALE: Pemetrexed may stop the growth of tumor cells by blocking some of the enzymes needed for their growth. Drugs used in chemotherapy, such as gemcitabine, work in different ways to stop the growth of tumor cells, either by killing the cells or by stopping them from dividing. Radiation therapy uses high energy x-rays to kill tumor cells.

PURPOSE: This phase I trial is studying the side effects and best dose of pemetrexed when given together with radiation therapy in treating patients with locally advanced pancreatic cancer.

DETAILED DESCRIPTION:
OBJECTIVES:

Primary

* Determine the maximum tolerated dose of pemetrexed disodium when given in combination with upper abdominal radiotherapy after induction therapy comprising gemcitabine hydrochloride and pemetrexed disodium followed by consolidation therapy with gemcitabine hydrochloride in patients with locally advanced pancreatic cancer.
* Determine the quantitative toxicity of this regimen in these patients.

Secondary

* Determine the quantitative and qualitative dose-limiting toxicities of pemetrexed disodium in combination with upper abdominal radiation therapy.
* Evaluate patterns of failure, response, and survival of these patients at 1 year

OUTLINE: This is an open-label, nonrandomized, dose-escalation study of pemetrexed disodium.

* Induction therapy: Patients receive pemetrexed disodium IV over 10 minutes and gemcitabine hydrochloride IV over 30 minutes on day 1. Treatment repeats every 14 days for 3 courses. Approximately 2 weeks later, patients without disease progression proceed to chemoradiotherapy.
* Chemoradiotherapy: Patients receive pemetrexed disodium IV over 10 minutes on days 1, 15, and 29 and undergo radiotherapy once daily 5 days a week for 5 ½ weeks. Approximately 2-3 weeks later, patients without disease progression proceed to consolidation therapy.

Cohorts of 3-9 patients receive escalating doses of pemetrexed disodium during chemoradiotherapy until the maximum tolerated dose (MTD) is determined. The MTD is defined as the dose at which ≤ 20% or ≤ 2 of 9 patients experience dose-limiting toxicity.

* Consolidation therapy: Patients receive gemcitabine hydrochloride IV over 30 minutes on days 1 and 8. Treatment repeats every 21 days for 2 courses in the absence of disease progression or unacceptable toxicity.

After completion of study treatment, patients are followed periodically.

PROJECTED ACCRUAL: A total of 25 patients will be accrued for this study.

ELIGIBILITY:
DISEASE CHARACTERISTICS:

* Histologically or cytologically confirmed carcinoma arising from the pancreas

  * Stage II or III disease, meeting 1 of the following criteria:

    * Nonresectable disease
    * Potentially resectable disease
    * Resectable disease
  * Stage IV disease with symptomatic back pain requiring palliation allowed at the discretion of the principal investigator
* Measurable, evaluable, or nonmeasurable disease
* No neuroendocrine tumor of the pancreas
* No documented brain metastasis
* No clinically significant pleural or peritoneal effusions that cannot be drained

PATIENT CHARACTERISTICS:

* ECOG performance status 0-1
* Life expectancy ≥ 12 weeks
* Absolute neutrophil count ≥ 1,500/mm³
* Platelet count ≥ 100,000/mm³
* Hemoglobin ≥ 9 g/dL
* Serum bilirubin ≤ 1.5 times upper limit of normal (ULN)
* Alkaline phosphatase ≤ 3 times ULN (5 times ULN if liver has tumor involvement)
* AST and ALT ≤ 3 times ULN (5 times ULN if liver has tumor involvement)
* Creatinine clearance ≥ 45 mL/min
* Not pregnant or nursing
* Negative pregnancy test
* Fertile patients must use effective contraception during and for 3 months after completion of study treatment
* No active infection
* No serious systemic disorders that would preclude study treatment
* No significant cardiovascular disease in the form of abnormal electrocardiogram coupled with clinical features of recent or recurrent cardiac disease (including myocardial infarction, angina, or hypertension)

PRIOR CONCURRENT THERAPY:

* More than 4 weeks since prior investigational agents
* No prior chemotherapy for pancreatic cancer
* Must be able to discontinue aspirin, dexamethasone, and other nonsteroidal anti-inflammatory agents for 2 days before, the day of, and 2 days after pemetrexed disodium dose (5 days before for long-acting agents such as piroxicam)
* Must be able and willing to take folic acid and cyanocobalamin (vitamin B12) supplementation

Ages: 18 Years to 120 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 4 (Actual)
Dates: Start 2005-10; Primary Completion 2008-05 (Actual); Study Completion 2008-05 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Arthur William Blackstock, MD, Study Chair — Wake Forest University Health Sciences
Locations (1):
- Wake Forest University Comprehensive Cancer Center, Winston-Salem, North Carolina, United States

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Pemetrexed in Combination With Concomitant Radiotherapy
Started | 4
Completed | 3
Not Completed | 1

BASELINE CHARACTERISTICS:
Arm/Group | Pemetrexed in Combination With Concomitant Radiotherapy
Number analyzed (Participants) | 4
Age, Continuous [Mean (Standard Deviation); unit: years] | 61.5 (2.645)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 2
  Male | 2

OUTCOME MEASURES:

1. Primary Outcome: Determine Maximum Tolerated Dose of Pemetrexed When Administered With Concomitant Radiation Therapy
Time Frame: 42 days
Population: data were not collected
Arm/Group | Pemetrexed in Combination With Concomitant Radiotherapy
Number analyzed (Participants) | 0

2. Primary Outcome: Quantitative Toxicity of Pemetrexed When Administered With Concomitant Radiation Therapy
Time Frame: 42 days
Population: data were not collected
Arm/Group | Pemetrexed in Combination With Concomitant Radiotherapy
Number analyzed (Participants) | 0

3. Secondary Outcome: Qualitative Dose-limiting Toxicities of Pemetrexed in Combination With Radiation Therapy
Description: Toxicity will be determined using the revised NCI Common Toxicity Criteria (CTC) version 3.0 for Toxicity and Adverse Event Reporting. Number of events with grade 1-5 will be reported.
Time Frame: 42 days
Population: Data available for 2 participants.
Measure: Number; unit: events
Arm/Group | Pemetrexed in Combination With Concomitant Radiotherapy
Number analyzed (Participants) | 2
events
  Grade 1 | 22
  Grade 2 | 7
  Grade 3 | 3
  Grade 4 | 0
  Grade 5 | 0

4. Secondary Outcome: Patterns of Failure
Time Frame: 1 year
Population: Data not collected.
Arm/Group | Pemetrexed in Combination With Concomitant Radiotherapy
Number analyzed (Participants) | 0

5. Secondary Outcome: Patterns of Response
Time Frame: 1 year
Population: Data not collected on all participants.
Measure: Count of Participants; unit: Participants
Arm/Group | Pemetrexed in Combination With Concomitant Radiotherapy
Number analyzed (Participants) | 3
Participants
  Partial Response | 1
  Stable disease | 2

6. Secondary Outcome: Number of Participants That Survived
Time Frame: 1 year
Measure: Count of Participants; unit: Participants
Arm/Group | Pemetrexed in Combination With Concomitant Radiotherapy
Number analyzed (Participants) | 3
Participants | 2

ADVERSE EVENTS:
Time Frame: up to 1 year
Arm/Group | Pemetrexed in Combination With Concomitant Radiotherapy
All-Cause Mortality (participants affected / at risk) | 1/4
Serious Adverse Events (participants affected / at risk) | 0/4
Other Adverse Events (participants affected / at risk) | 2/4
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Pemetrexed in Combination With Concomitant Radiotherapy (N=4)
ALT, SGPT (Gastrointestinal disorders) | 1 — serum glutamic pyruvic transaminase
Alkaline phosphatase (Gastrointestinal disorders) | 1
Anorexia (Gastrointestinal disorders) | 1
Calcium, serum-high (Blood and lymphatic system disorders) | 1 — hypercalcemia
Calcium, serum-low (Blood and lymphatic system disorders) | 1 — hypocalcemia
Constipation (Gastrointestinal disorders) | 2
Dehydration (Renal and urinary disorders) | 1
Dizziness (General disorders) | 1
Edema (Skin and subcutaneous tissue disorders) | 1 — limb
Edema (Skin and subcutaneous tissue disorders) | 1 — trunk/genital
Fatigue (General disorders) | 1 — asthenia, lethargy, malaise
Fever (in the absence of neutropenia, where neutropenia is defined as ANC <1.0 x 10e9/L) (General disorders) | 1 — in the absence of neutropenia, where neutropenia is defined as ANC <1.0 x 10e9/L
Gastrointestinal - Other (Gastrointestinal disorders) | 2
Glucose, serum-high (Metabolism and nutrition disorders) | 2 — hyperglycemia
Glucose, serum-low (Metabolism and nutrition disorders) | 1 — hypoglycemia
Hemoglobin (gender based) (Blood and lymphatic system disorders) | 2
Infection - Other (Infections and infestations) | 1
Infection with normal ANC or Grade 1 or 2 neutrophils (Infections and infestations) | 1 — Penis
Leukocytes (total WBC) (4.8-10.8) (Blood and lymphatic system disorders) | 2
Nausea (Gastrointestinal disorders) | 1
Neurology - Other (Nervous system disorders) | 1
Neuropathy (Nervous system disorders) | 1 — sensory
Neutrophils/granulocytes (ANC/AGC) 1.6-7.3 (Immune system disorders) | 2
Ocular/Visual - Other (Eye disorders) | 1
Pain - Other (General disorders) | 1
Pain (Gastrointestinal disorders) | 1 — Stomach
Platelets (Blood and lymphatic system disorders) | 1 — (160-360)
Potassium, serum-high (Blood and lymphatic system disorders) | 1 — (hyperkalemia) (3.5-5.3)
Rash (Skin and subcutaneous tissue disorders) | 1 — dermatitis associated with radiation
Renal/Genitourinary - Other (Renal and urinary disorders) | 1
Sodium, serum-high (Renal and urinary disorders) | 1 — (hypernatremia) (135-146)
Watery eye (Eye disorders) | 1 — (epiphora, tearing)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes